CLINICAL TRIAL: NCT07079995
Title: Healthy School Recognized Campus: A Hybrid Type 2 Implementation-Effectiveness Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HSRC DRCT STUDY2025-0650
Record Dates: First submitted 2025-07-01; First posted 2025-07-23 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases; Physical Activity; Nutrition
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity | interventions — Waiting Lists

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HSRC + Standard Implementation (No Intervention): Participants in this group will receive HSRC in the first year of enrollment with standard implementation. [schools (n=5), participants (n=225)]
- HSRC + Mentoring Program (Experimental): Participants in this group will receive HSRC in the first year of enrollment with the mentoring program. [schools (n=5), participants (n=225)]
  Interventions: Behavioral: Mentoring program
- Waitlist Control + HSRC + Standard Implementation (Experimental): Participants in this group will receive HSRC with standard implementation one year after enrollment. [schools (n=5), participants (n=225)]
  Interventions: Behavioral: Waitlist
- Waitlist Control + HSRC + Mentoring Program (Experimental): Participants in this group will receive HSRC with the mentoring program one year after enrollment. [schools (n=5), participants (n=225)]
  Interventions: Behavioral: Mentoring program; Behavioral: Waitlist

INTERVENTIONS:
Behavioral: Mentoring program — Schools in this group will participate in meetings and receive newsletters to help with program implementation.
  Arms: HSRC + Mentoring Program; Waitlist Control + HSRC + Mentoring Program
Behavioral: Waitlist — Schools in this group will wait 1 year to receive HSRC. Schools will not add or remove any current physical activity and/or healthy eating programs.
  Arms: Waitlist Control + HSRC + Mentoring Program; Waitlist Control + HSRC + Standard Implementation

SUMMARY:
Healthy School Recognized Campus is a Texas A&M AgriLife Extension initiative that supports the delivery of school-based physical activity and nutrition programs for diverse youth across Texas. The purpose of this study is to conduct a type 2 hybrid implementation-effectiveness, cluster dual randomized controlled trial (DRCT) to assess both Healthy School Recognized Campus (HSRC) and the mentoring program.

DETAILED DESCRIPTION:
This study uses a type 2 hybrid implementation-effectiveness, cluster dual randomized controlled trial (DRCT). DRCTs include two randomized controlled trials within the same study: one testing an intervention (i.e., HSRC) and one testing an implementation strategy (i.e., the mentoring program).

Schools in Central and East Texas (n=20) of similar socio-economic status will be randomized at baseline to either the HSRC condition or the Waitlist Control condition. In the HSRC condition, schools will attempt to deliver youth and adult physical activity or nutrition programs. In the Waitlist Control condition, schools will not add or remove any current physical activity and/or healthy eating programs, and will receive HSRC the next school year. Schools will also be randomized to receive the mentoring program or standard implementation immediately or after being a waitlist control.

Aim 1: Determine the effectiveness of the HSRC initiative compared to a control group on BMI-Z score, physical activity, and skin carotenoids (i.e., fruit and vegetable intake).

For Aim 1, the investigators will compare outcomes in 10 Texas schools that receive HSRC with 10 Waitlist Control communities.

Aim 2: Determine the impact of the mentoring program compared to standard implementation on short-term (acceptability, appropriateness, feasibility) and long-term (number of students reached, total dosage delivered) implementation outcomes.

For Aim 2, the investigators will compare outcomes in 10 Texas schools that receive the mentoring program with 10 that receive standard implementation.

ELIGIBILITY:
School Inclusion Criteria:

* located in Central and East Texas
* Public school

Student Inclusion Criteria

* enrolled in the 4th, 5th, 6th, 7th, 8th, or 9th grade
* able to read, speak, and write in English

Student Exclusion Criteria:

* any motor or cognitive impairments or other health conditions that would prevent them from completing a physical assessment

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Body mass index (BMI) | Baseline, 9 months
  Weight will be measured with a scale (in pounds), and height will be measured using a stadiometer (in inches). Weight and height will be combined to report BMI as follows, BMI = (weight (lb)/height (inches)2) x 703.
Acceptability of the HSRC program | Baseline, 9 months
  Acceptability will be assessed using the Acceptability of Intervention Measure (AIM) 4-item survey. The survey will be used to assess program implementers' perceived acceptability of the program (i.e., This program seems fine.)
Appropriateness of the HSRC program | Baseline, 9 months
  Appropriateness will be assessed with the Intervention Appropriateness Measure (IAM) 4-item survey. The survey will assess program implementers' perception of the appropriateness of the program (e.g., This program seems suitable.)
Feasibility of the HSRC program | Baseline, 9 months
  Feasibility will be assessed using the Feasibility of Intervention Measure (FIM) 4-item survey. The survey will assess program implementers' perception of the program's feasibility (e.g., This program seems doable.)

SECONDARY OUTCOMES:
Concentration of subdermal carotenoids | Baseline, 9 months
  The concentration of subdermal carotenoids will assess the changes in fruit and vegetable consumption using the Veggie Meter: A non-invasive, portable machine that measures subdermal carotenoid levels using resonance Raman spectroscopy.
Accelerometer-derived physical activity estimation | Baseline, 9 months
  Physical activity will be measured using Actigraph accelerometers. Measurements will include light physical activity (PA), moderate PA, moderate to vigorous PA, and vigorous PA.
Number of students reached | Baseline, 9 months
Total program dosage delivered | Baseline, 9 months

OTHER OUTCOMES:
Blood pressure | Baseline, 9 months
  Blood pressure (systolic and diastolic) will be measured with two numbers using an automated Omron sphygmomanometer.
Physical fitness capacity estimation | Baseline, 9 months
  Physical fitness will be measured using the FitnessGram PACER multistage aerobic capacity test: Children will run back and forth 20 meters, with an initial running speed of 8.5 km/hour and a progressive 0.5-km/hour increase in running speed every minute. As the test continues it becomes progressively harder. The number of laps completed is used to estimate children's physical fitness physical fitness.
Waist circumference | Baseline, 9 months
  Waist circumference will be measured at the midpoint between the floating rib and iliac crest using a tape measure.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Szeszulski, Principal Investigator — Institute for Advancing Health through Agriculture
Locations (1):
- Texas A&M AgriLife Dallas Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will include student biometrics, student surveys, and implementer surveys. Student biometrics will include assessments of height, weight, physical activity, fruit and vegetable consumption, cardiovascular fitness, and markers of cardiometabolic health (e.g., blood pressure). Student surveys will include assessment of student demographics, physical activity, healthy eating, and other important outcomes (e.g., positive youth development). Implementer surveys will include demographics and assessment of implementation outcomes as they relate to programs that are a part of healthy school recognized campus.
Time Frame: start: 3/31/2028
Access Criteria: Researchers can access through ClinicalTrials.gov or Open Science Framework (general)

REFERENCES:
- [Derived] Schaefers A, Beattie CM, de Mello GT, George A, Marstall K, Gardner J, Szeszulski J. Healthy school recognized campus: design and methodology of a hybrid type 2 implementation-effectiveness cluster randomized trial. Implement Sci. 2026 Feb 5. doi: 10.1186/s13012-026-01487-2. Online ahead of print. PMID 41645239